CLINICAL TRIAL: NCT00625742
Title: An Exploratory Trial of a Multimodal Treatment Strategy for Cancer Cachexia
Brief Title: Multimodal Treatment Strategy for Cancer Cachexia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0739; NCI-2012-01744 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-01

CONDITIONS: Advanced Cancer; Cachexia
Keywords: Advanced Cancer; Cancer Cachexia; Cachexia; Melatonin; Juven; Exercise Training; Weight Loss
MeSH Terms: conditions — Cachexia; Weight Loss | interventions — Exercise; Melatonin; Atenolol; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multimodal Treatment Strategy (Experimental): Exercise Program + Pharmacologic Intervention (Melatonin + Atenolol + Ibuprofen) + Nutritional Supplementation (Juven) - Resistance training sessions twice weekly using Thera-bands. Walking or running for 3-4 minutes at 70-80% of maximum predicted heart rate. Melatonin 20 mg by mouth (PO) Daily. 90 calories of Juven, twice a day.
  Interventions: Behavioral: Graded Resistance Training; Behavioral: Aerobic Exercise; Drug: Melatonin; Dietary Supplement: Juven; Drug: Atenolol; Drug: Ibuprofen

INTERVENTIONS:
Behavioral: Graded Resistance Training — Resistance training sessions twice weekly using Thera-bands.
Behavioral: Aerobic Exercise — Walking or running for 3-4 minutes at 70-80% of your maximum predicted heart rate.
Drug: Melatonin — 20 mg by mouth (PO) Daily
Dietary Supplement: Juven — 90 calories of Juven, twice a day.
Drug: Atenolol — Atenolol will only be taken if there's evidence of increased sympathetic activity (resting heart rate >110 beats/min) or resting energy expenditure (REE) > 110% of predicted.
Drug: Ibuprofen — Ibuprofen 1200mg/day in three divided doses.

SUMMARY:
The primary aim of this proposal is to present a novel, multimodal treatment strategy for increasing lean body mass in individuals with cancer who experience cachexia between baseline and day 29 (+/- 3 days). The strategy includes graded resistance training and aerobic exercise, targeted nutrient supplementation and pharmacologic intervention (melatonin).

We postulate that this strategy, together with the simultaneous management of symptoms that decrease appetite (e.g. depression, pain, and nausea), will also accomplish our secondary objectives of improving clinical outcomes such as strength and function between baseline and day 29 (+/- 3 days).

DETAILED DESCRIPTION:
The Study Drugs:

Melatonin is a hormone that helps reduce inflammation and poor food absorption caused by cancer. It may also enhance the effects of ibuprofen.

Juven is a nutritional supplement that is designed to help build muscle and slow muscle breakdown.

Screening Tests:

Before you can start treatment on this study, you will have "screening tests" to help the doctor decide if you are eligible to take part in this study. The following tests will be performed:

* Blood (1 to 2 tablespoons) will be drawn for routine tests. This routine blood draw will include a pregnancy test for women who are able to have children. To be eligible to take part in this study, the pregnancy test must be negative.
* Additional blood (1 tablespoon) will be drawn to check your thyroid function and the levels of two B vitamins, if these have not been checked within the past 3 months.
* You will have a physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate).
* You will have an electrocardiogram (ECG -- a test that measures the electrical activity of the heart).
* Your resting energy expenditure (energy used at rest) will be measured. with a calorie-measuring device. For this test, you will breathe in and out through your mouth for about 10 minutes to allow a calorie-measuring device to measure the oxygen your body uses, and from this it calculates how much energy your body uses at rest.
* You will be asked to fill out a questionnaire to rate your overall physical well-being, another questionnaire to rate your level of fatigue, and a third questionnaire to rate your experiences with 10 common symptoms in the past 24 hours (pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, changes in appetite, sleep difficulty, and feeling of well being). In total, these questionnaires will take about 30 minutes to complete.
* You will complete a diary entry that lists all of the food and drinks you have had in the last 3 days. It should take about 10 minutes to complete.
* Your strength and stamina will be evaluated. This is measured by hand-grip and pinch strength tests that are done with both hands. These tests will see how hard you can grip a device with your hand and pinch the pads of another device called a pinch gauge. These tests will be done 3 times and your best scores will be used. Your strength and stamina will also be checked using the Get-Up-and-Go test and the 6-minute walk test. The Get-Up-and-Go test measures how long it takes to get up from sitting in a chair that has arms, walking 10 feet, turning around and walking back to the chair, and sitting down. The 6-minute walk test will measure the distance you can walk in 6 minutes on a 100-foot loop. You will walk 50 feet and then turn and walk back to the beginning. You will do this at a walking speed that feels comfortable and for as many times as you can in 6 minutes.
* Blood (1 to 2 tablespoons) will be drawn to check for markers of inflammation and nutrition status.

Study Drug Administration:

You will take one (1) 20mg capsule of melatonin every night. It can be taken with or without food. It should be taken with 8 ounces (1 cup) of water.

You will drink 90 calories of Juven, twice a day. Juven is a powder supplement that is mixed into 8 ounces of water. It is available in orange or grape flavors.

You will also be instructed to increase your daily calorie intake by at least 1,000 calories. To assist you in doing so, dietary advice will be given to you by a nurse or physician.

Exercise Training:

You will complete 2 exercise training sessions a week. The sessions will combine resistance and graded aerobic training.

Resistance training (with Thera-bands) is designed to increase the muscle-building effects of a hormone called testosterone. Thera-bands are rubber bands that you can hold or put around your feet to provide resistance to your muscles when you bend and flex your arms and legs.

You will be instructed in how to do 3 upper-body exercises (chest press, shoulder press, and arm pull down) and 3 lower-body exercises (leg press, leg extension, and leg flexion).

At your first visit, a physician will educate you to make sure that all exercises are done correctly.

Each repetition will take 12 seconds to complete (6 seconds to bend, then 6 seconds to straighten your arm or leg). When 6 repetitions are completed, the next week's set will be increased by 1 repetition.

Graded aerobic exercise is a walking/running program that may help you exercise longer.

Graded aerobic exercise involves walking or running for 3-4 minutes at 70-80% of your maximum predicted heart rate. There will be a 3-minute warm-up and a 3-minute cool-down before and after this exercise.

During your first visit, you will be shown how to monitor your heart rate and how to exercise at 70-80% of your maximum heart rate.

You will add 1 minute to your aerobic exercise at the start of each week.

You will receive your own customized aerobic and resistance exercise program based on your range of motion and risk for falls, which will be evaluated by the study staff.

If you experience chest pain, have a temperature over 100.4 °F, have a platelet count of lower than a certain level, have fresh bruises, or shortness of breath at rest, you will be advised to stop exercising until these are relieved.

Evaluations:

While on study, within 3 days of the days listed below, the following measurements will be monitored:

* Your lean body mass and weight will be checked at Days 15 and 29 using the Tanita TBF-310 body composition analyzer/scale. For measurements with the Tanita TBF 310, you will be asked to wear light clothes and to take off your shoes and socks when being weighed. You will stand on a special scale that will send an extremely low-energy, high-frequency electrical signal from one foot to your other foot. You should not be able to feel this at all.
* Your muscle mass (mid-arm muscle area) will be measured with a special tape.
* The thickness of a skin fold on your triceps (back of your upper arm) will be measured 3 times using skin fold calipers. Calipers are a gentle clamp-like device that is used on the outside of your body to measure skin thickness.
* At Day 29, your resting energy expenditure will be measured.
* On Days 15 and 29 of the study cycle, you will complete the same 3 questionnaires as at screening.
* Your caloric intake will be measured on Days 15 and 29.
* Your strength and stamina will be evaluated on Days 15 and 29.
* On Day 29, blood (1 to 2 tablespoons) will be drawn to check for markers of inflammation and nutrition.
* Blood (about 1 to 2 tablespoons) will be drawn for routine tests every 15 days while you are on-study. You will also have a fecal occult blood test at this time.

Length of Study:

You will be on study for 29 days (1 cycle).

This is an investigational study. Melatonin and Juven are commercially available nutritional supplements and are exempt from FDA approval. However, in patients with cancer and cachexia, the study treatment (resistance training, aerobic exercise, and the use of Juven, and melatonin) is considered experimental. At this time, it is only being used in research.

Up to 40 patients will be enrolled on this study. Up to 30 patients will be enrolled at M.D. Anderson, and 10 will be enrolled at the University of Alabama-Birmingham.

ELIGIBILITY:
Inclusion Criteria:

1. Are referred to the Cachexia Clinic with involuntary weight loss of >5% of their premorbid weight within the previous 6 months.
2. Are 18 years of age or older
3. Have a Karnofsky performance score of 60 or higher.
4. Can maintain oral food intake during the study
5. Can understand the study procedures and can sign an informed consent form.
6. Are not currently taking melatonin.
7. Are taking megestrol acetate and continue to lose weight despite at least 2 weeks of therapy.
8. Have a calculated creatinine clearance of >/= 60 cc/min.

Exclusion Criteria:

1. Have dementia or delirium (as determined by the palliative care specialist) at study entry.
2. Are pregnant
3. Have been taking corticosteroids for longer than 48 hours.
4. Have pulmonary edema, ascites or pitting edema on clinical examination.
5. Are unable to walk.
6. Have a history of serious adverse gastrointestinal events (i.e., bleeding or perforation),history of a coagulopathy or current anti-coagulant use.
7. Have an ALT/AST>3x upper limit of normal.
8. Patients on methotrexate.
9. Patients taking melatonin receptor agonists (such as Rozerem® [ramelteon]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rony Dev, DO, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 18, 2008 to December 15, 2010. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Early termination of the study due to follow-up issues and low recruitment numbers.
Groups:
- Multimodal Treatment Strategy: Exercise Program + Pharmacologic Intervention (Atenolol + Ibuprofen + Melatonin) + Nutritional Supplementation (Juven) - Resistance training sessions twice weekly using Thera-bands. Walking or running for 3-4 minutes, and Oral Melatonin 20 mg Daily. 90 calories of Juven, twice a day.
Period: Overall Study
Arm/Group | Multimodal Treatment Strategy
Started | 15
Completed | 3
Not Completed | 12
Not completed — Disease Progression | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 4
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Multimodal Treatment Strategy
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 57 [34 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Participant Gain in Lean Body Mass
Description: Measure increases in lean body mass in individuals with cancer who experience cachexia between baseline and day 29 (+/- 3 days).
Time Frame: Baseline to Day 29, approximately 30 days
Population: Only 3 patients completed the study and were evaluable for analysis, others were unable to follow the study exercise and intervention elements. There were insufficient data points collected to analyze.
Arm/Group | Multimodal Treatment Strategy
Number analyzed (Participants) | 0

2. Secondary Outcome: Improvement of Clinical Outcomes
Description: Improvement of clinical outcomes such as strength and function between baseline and day 29 (+/- 3 days).
Time Frame: Baseline to Day 29, approximately 30 days
Population: as for outcome 1
Arm/Group | Multimodal Treatment Strategy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collection from baseline to day 29 (+/- 3 days). Overall collection period: October 24, 2008 to January 24, 2011.
Arm/Group | Multimodal Treatment Strategy
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multimodal Treatment Strategy (N=15)
Dizziness (Nervous system disorders) | 1 (1)
Dry Mouth (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 2 (2)
Cord Compression (Musculoskeletal and connective tissue disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multimodal Treatment Strategy (N=15)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
Anxiety (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (8)
Depressed level of consciousness (Nervous system disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4)
Dry mouth (General disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 9 (9)
Headache (Nervous system disorders) | 1 (1)
Hemorrhage nasal (Vascular disorders) | 1 (1)
Insomnia (Nervous system disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (6)
Neurology (Other) (Nervous system disorders) | 1 (1)
Oral pain (General disorders) | 2 (2)
Pain, Muscle (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (Other) (General disorders) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope vasovagal (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The sample size of the available data is too small to detect any significant differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes